CLINICAL TRIAL: NCT05023564
Title: Peking Union Medical College Hospital (PUMCH) Dementia Longitudinal Cohort Study
Brief Title: PUMCH Dementia Longitudinal Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH Dementia Cohort
Record Dates: First submitted 2021-07-31; First posted 2021-08-26 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Dementia; Dementia, Vascular; Dementia With Lewy Bodies; Dementia, Mixed; Dementia Alzheimers; Dementia Frontal; Dementia, Mild
MeSH Terms: conditions — Dementia; Dementia, Vascular; Lewy Body Disease; Mixed Dementias; Alzheimer Disease; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, CSF,urine,skin tissue, brain tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early onset dementia: Dementia patients with onset age lower than 65y/o
- Late onset dementia: Dementia patients with onset age between 65y/o and 85y/o
- Oldest old dementia: Dementia patients with onset age older than 85y/o
- Cognitive normal control: Normal Aging with normal cognitive function

SUMMARY:
The PUMCH Dementia Cohort is a hospital-based, observational study of Chinese elderly with cognitive impairment.

DETAILED DESCRIPTION:
In China, the burden of dementia is increasing, which has a major impact on medical care, society, and the economy. In order to solve this important public health problem, a cohort study of cognitive impairment in the elderly should be carried out. We designed an age stratified dementia cohort and tried to to clarify the risk and prognostic factors, disease characteristics, cognitive evaluation, biomarkers, diagnosis, treatment of dementia and its subtypes in China. It is of great significance to establish a relatively comprehensive dementia database, improve the level of clinical diagnosis and treatment of cognitive impairment, and formulate prevention and treatment strategies for dementia.

Baseline data collection and cohort establishing: Detailed clinical information including demographic data, clinical history, past history and physical examination are collected. Formatted neuropsychological battery is used in all patients, including screening tests (MMSE, MoCA-PUMCH, ADL, HAD) and domain specific evaluation (Memory, executive function, visual spatial, calculation, language). Samples including serum, CSF, urine, skin, saliva are stored. Every patient is followed up every 6 months. Autopsy brain tissue will be collected if patients died.

The main contents of this study are following:

1. Explore the relationship between lifestyles, stress and dementia.
2. Assess risk factors for dementia.
3. Evaluating behavioral and psychological symptoms of dementia.
4. Improve the long-term follow-up cohort stratified by age and dementia type and construct the high standard information and sample bank.
5. Explore biomarkers of different groups of dementia, incorporating neuropsychology, multi-model neuroimaging, metabolics and proteomics based fluid biomarkers as well as genetic biomarkers. Autopsy after clinical follow up help to verify the biomarkers.
6. Establish and promote standardized and consistent biomarker detection methods.
7. Dementia education and training.
8. Use machine learning methods to establish computer-assisted dementia diagnosis system and evaluation system. Establish prediction models for the progression of dementia.

ELIGIBILITY:
Inclusion Criteria:

* Neurodegenerative dementia diagnosis based on 2011 NIA-AA criteria of Dementia
* Fixed care giver and can follow up regularly

Exclusion Criteria:

* Not demented, including MCI
* Systemic severe diseases and severe vision or hearing problem effecting follow up and neuropsychological evaluation
* Without fixed care giver
* Reject informed consent
* Expected life shorter than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We included age stratified dementia (early onset, late onset, oldest old) , including AD, FTD,VaD, DLB and mixed dementia. Also we include cognitive normal controls.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of dementia | Through study completion,an average of 10-20 years
  Through follow up of cognitive normal control ,to find the incidence of dementia in PUMCH cohort
The relationship between lifestyles, stress (stressful events and their degree) and dementia | Through study completion,an average of 10 years
  Analysis of the relationship between lifestyles, stress and progression of dementia. Discover lifestyle factors (such as diet, residential environment, physical activity, hobbies, and sleep) and stress (stressful events and their degree) by using a questionnaire designed by PUMCH
Risk factors for dementia | Through study completion,an average of 10-20 years
  Collect the risk factors in normal control and analysis the relationship after diagnosis of dementia
Cognitive decline | Through study completion,an average of 10-20 years
  Use a systematic neuropsychological battery designed by PUMCH
Functional decline | Through study completion,an average of 10-20 years
  Use Activity of Daily Living Scale（ADL）
Changes in the Neuropsychiatric Index (NPI) | Through study completion,an average of 10 years
  In dementia patients, analysis their behavioral and psychological symptoms and the related factor. Discover the relationship between behavioral and psychological symptoms and biomarkers for dementia.
Changes in the Hospital Anxiety and Depression scale (HAD) | Through study completion,an average of 10 years
  In dementia patients, analysis their behavioral and psychological symptoms and the related factor. Discover the relationship between behavioral and psychological symptoms and biomarkers for dementia.
Changes in the Cornell Scale for dementia | Through study completion,an average of 10 years
  In dementia patients, analysis their behavioral and psychological symptoms and the related factor. Discover the relationship between behavioral and psychological symptoms and biomarkers for dementia.
Tau and Beta-amyloid biomarkers in CSF | Through study completion,an average of 10 years
  Concentration ( pg/mL) of beta-amyloid, tau and phospho-tau in cerebrospinal fluid (CSF) of patients with dementia and controls
Tau biomarkers in serum | Through study completion,an average of 10 years
  Concentration ( pg/mL) of tau in serum of patients with dementia and controls
CSF collection for assessing new dementia biomarker | Through study completion,an average of 10 years
  Use collected CSF to assess new biomarkers.
Serum collection for assessing new dementia biomarker | Through study completion,an average of 10 years
  Use collected serum to assess new biomarkers.
Urine collection for assessing new dementia biomarker | Through study completion,an average of 10 years
  Use collected urine to assess new biomarkers.
Skin collection for assessing new dementia biomarker | Through study completion,an average of 10 years
  Use collected skin for finding new biomarkers.
Biomarker differences of dementia | Through study completion,an average of 10 years
  The differences of biomarkers in patients with different dementia.
Incorporating age stratified biomarkers into the diagnosis of dementia | Through study completion,an average of 10 years
  Comparing the relationships between biomarkers and clinical presentations. Incorporate biomarkers into the accurate and early diagnosis of dementia
Dementia education and training | Through study completion,an average of 10 years
  Observe the function of education and training in the treatment and care of dementia patients
Dementia diagnosis system and evaluation system | Through study completion,an average of 10 years
  Use machine learning methods to establish computer-assisted dementia diagnosis system and evaluation system. Establish prediction models for the progression of dementia

CONTACTS AND LOCATIONS:
Overall Officials: Chenhui Mao, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] Olsson B, Lautner R, Andreasson U, Ohrfelt A, Portelius E, Bjerke M, Holtta M, Rosen C, Olsson C, Strobel G, Wu E, Dakin K, Petzold M, Blennow K, Zetterberg H. CSF and blood biomarkers for the diagnosis of Alzheimer's disease: a systematic review and meta-analysis. Lancet Neurol. 2016 Jun;15(7):673-684. doi: 10.1016/S1474-4422(16)00070-3. Epub 2016 Apr 8. PMID 27068280
- [Background] Norton S, Matthews FE, Barnes DE, Yaffe K, Brayne C. Potential for primary prevention of Alzheimer's disease: an analysis of population-based data. Lancet Neurol. 2014 Aug;13(8):788-94. doi: 10.1016/S1474-4422(14)70136-X. PMID 25030513
- [Background] McKhann GM, Albert MS, Grossman M, Miller B, Dickson D, Trojanowski JQ; Work Group on Frontotemporal Dementia and Pick's Disease. Clinical and pathological diagnosis of frontotemporal dementia: report of the Work Group on Frontotemporal Dementia and Pick's Disease. Arch Neurol. 2001 Nov;58(11):1803-9. doi: 10.1001/archneur.58.11.1803. PMID 11708987
- [Background] Rosenberg A, Ngandu T, Rusanen M, Antikainen R, Backman L, Havulinna S, Hanninen T, Laatikainen T, Lehtisalo J, Levalahti E, Lindstrom J, Paajanen T, Peltonen M, Soininen H, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Solomon A, Kivipelto M. Multidomain lifestyle intervention benefits a large elderly population at risk for cognitive decline and dementia regardless of baseline characteristics: The FINGER trial. Alzheimers Dement. 2018 Mar;14(3):263-270. doi: 10.1016/j.jalz.2017.09.006. Epub 2017 Oct 19. PMID 29055814
- [Derived] Yang X, Wu M, Liang M, Zhang H, Li B, Mao C, Dong L, Wang Y, Xing H, Ren C, Huang Z, Wen Q, Ge Q, Yu Z, Feng F, Gao J, Huo L. Ultra-fast [18F]florbetapir PET imaging using the uMI Panorama PET/CT system. EJNMMI Phys. 2024 Dec 30;11(1):107. doi: 10.1186/s40658-024-00712-5. PMID 39738784